CLINICAL TRIAL: NCT05003076
Title: Drug Effects on EEG
Brief Title: Brain Function and EEG
Acronym: DEG
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB21-0769
Record Dates: First submitted 2021-08-06; First posted 2021-08-12 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Healthy; Mood
MeSH Terms: interventions — Methamphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Then Methamphetamine (Experimental): Participants first receive placebo at their first session in the laboratory. Then will return to the laboratory 72 hours later and will receive 20 mg methamphetamine.
  Interventions: Drug: Methamphetamine; Drug: Placebo
- Methamphetamine Then Placebo (Experimental): Participants first receive 20 mg methamphetamine at their first session in the laboratory Then will return to the laboratory 72 hours later and will receive placebo.
  Interventions: Drug: Methamphetamine; Drug: Placebo

INTERVENTIONS:
Drug: Methamphetamine — Participants will be given 20 mg of Methamphetamine.
Drug: Placebo — Participants will be given a placebo capsule that will only contain lactose.

SUMMARY:
In this project, we will examine effects of MA on reward function using electroencephalograms (EEG), which will complement our ongoing study with MA and fMRI. We will determine how MA alters reward-related neural activity and how this is related to its subjective rewarding effects. The effects of MA on reward function will be examined using both reward-task-related activation and resting state activity. We will examine the effects of MA on ratings of drug liking and euphoria, as well as on EEG measures sensitivity to reward. Healthy young adults will undergo three EEG sessions with placebo and MA (10 and 20 mg), while performing the Monetary Incentive Delay task and the Stop Task, as a measure of inhibition. We will examine correlations between the neural responses and subjective responses to MA.

Our central hypotheses are 1) that MA will increase feelings of alertness and well-being, and 2) that MA will increase neural responses to anticipation and receipt of reward, and 3) that the effects of MA on mood will be correlated with its effects on neural responses to reward.

ELIGIBILITY:
Inclusion Criteria:

BMI between 19 and 26 Less than 4 alcohol or caffeinated beverages a day.

Exclusion Criteria:

High blood pressure

Any medical condition requiring regular medication Individuals with a current (within the last year) DSM-IV Axis 1 diagnosis Individuals with a history of dependence on stimulant drugs Women who are pregnant or trying to become pregnant.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Change in SUbjective Effects as Assessed by Score on "Feel Drug", "Feel High", "Like Drug", and "Want More" Sub-scales of Drug Effects Questionnaire (DEQ). | Time Frame: Day 1(baseline), 3
  Participants will complete The Drug Effects Questionnaire during the initial baseline session to determine their subjective stimulant profile. The Dug Effects Questionnaire (DEQ) is a visual analog scale questionnaire that assesses the extent to which subjects experience four subjective states: "Feel Drug", "Feel High", "Like Drug", and "Want More". All sub-scales are scored on a visual analogue scale (Scroll bar on computer screen) ranging from 0-100. 100 represents the highest score for that subjective state, and the higher the score, the worse the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Harriet de Wit, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No